CLINICAL TRIAL: NCT00900003
Title: Developing Biomarkers in Pancreatic Cancer
Brief Title: Studying Biomarkers in Patients With Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Associate Professor; Radiation Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC GI 0717; P30CA068485 (NIH); VU-VICC-GI-0717; VU-VICC-070366
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pancreatic cancer patients: pancreatic cancer patients with excess tissue collected at the time of standard of care surgery
  Interventions: Genetic: protein analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: protein analysis — Using material that is already being acquired as a component of clinical care (only that which is excess after routine clinical care), we will determine if pre-treatment markers can be used to correlate with clinical outcomes of survival and recurrence. Examples of such markers include studying if the integrity of DNA repair pathway in pancreatic cancers, analyzed by Rad51 and phosphorylated DNA-PK foci formation, correlates with tumor response to radiotherapy, chemotherapy, and overall survival. The markers targeted are proteins secreted by cancer cells and/or cancer associated cells.
Other: laboratory biomarker analysis — A method of extracting and identifying secreted cytokines and growth factors from tissues of the quantity of typical biopsy tissues has been developed.The purpose of this study is to determine if this method of biomarker discovery can now be applied to pancreatic cancer population.

SUMMARY:
RATIONALE: Studying samples of tissue in the laboratory from patients with cancer may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in patients with pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether the cellular localization of BRCA1 can predict how patients with pancreatic cancer will respond to cytotoxic agents (e.g., fluorouracil or gemcitabine hydrochloride) or radiotherapy.
* To identify pre-treatment markers that can be used to correlate with clinical outcomes of survival and recurrence.
* To determine if a method of extracting and identifying secreted cytokines and growth factors from biopsy tissue can now be applied to the pancreatic cancer population.

OUTLINE: Tissue samples from biopsies performed during pancreatectomy are collected from the Vanderbilt Ingram Cancer Center Human Tissue Acquisition Core for laboratory biomarker studies. Proteins secreted by cancer cells and/or cancer-associated cells are studied by extracting and identifying secreted cytokines and growth factors from biopsy tissue. The integrity of the DNA repair pathway in pancreatic cancer is analyzed by Rad51 and phosphorylated DNA-PK foci formation. Markers are correlated with clinical outcome.

Patients are followed for recurrence, relapse, and death from disease.

ELIGIBILITY:
Inclusion criteria

* Any subject with excess tissue collected at time of routine surgery for pancreatic cancer is eligible.
* All subjects participating in this protocol will be followed for recurrence, relapse and death from disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with cancer of the pancreas
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2007-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cellular localization of BRCA1 as a predictor of response to cytotoxic agents or radiotherapy | following collection of all pancreatic tissue specimens and patient outcome data
  Examine the location of BRCA1 in the cells and determine if this location predicts patient response to the chemotherapy drugs given

SECONDARY OUTCOMES:
Correlation of pre-treatment markers with survival and recurrence | at expiration date of final patient enrolled
  Compare and contract of biomarkers in patient's tissue that are detected before treatment has a relationship to their survival and recurrence of their cancer
Application of a method of extracting and identifying secreted cytokines and growth factors from biopsy tissue to the pancreatic cancer population | upon collection of pancreatic tissue for each patient
  Researchers will determine if the methods they have developed for extracting and identifying cytokines in biopsy tissue can be applied to the pancreatic cancer tissue

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/